CLINICAL TRIAL: NCT05654428
Title: Effects of Mackenzie Extension and William Flexion Exercises in Lumbo-Sarcal Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Collaborators: National Institute of Rehabilitation Medicine, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, Muhammad salman, PT, Principal researcher, Isra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 337
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Lumbosacral Radiculopathy

STUDY DESIGN:
Intervention Model Description: A Randomized Control Trail with 2 Equal groups
Who Masked: Participant
Masking Description: Just Participants are unaware about which type of intervention they are being underwent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): 55 patients
  Standard treatment:
  TENS (4-pole) + Hot pack for 15 minutes Standard treatment:
  TENS (4-pole) + Hot pack for 15 minutes
  New Intervention:
  Mckenzie Extension
  * Prone press-ups
  * Head life in prone
  * Prone on elbow
  * Prone on hands
  * Prone on pillow
  Interventions: Other: Mckenzie Extension Exercises
- Control Group (Active Comparator): 55 patients
  Standard treatment:
  TENS (4-pole) + Hot pack for 15 minutes Standard treatment:
  TENS (4-pole) + Hot pack for 15 minutes
  New Intervention:
  William Flexion
  * Single knee to chest
  * Double knee to chest
  * Straight Leg Raise
  * Bridging
  * Pelvic tilt
  Interventions: Other: William Flexion Exercises

INTERVENTIONS:
Other: Mckenzie Extension Exercises — The exercises used to create space between under lying structures of lumber spine which help centralization of pain and can be performed in prone lying such as prone press ups, prone on elbow, and head lift in prone.
  Arms: Experimental Group
Other: William Flexion Exercises — Exercises for strengthening of gluteal and abdominal muscles which help to reduce pressure on the nerve root by promoting flexion at lumber spine such as knee to chest, double knee to chest, bridging(Gluets bridge), and straight leg raise (SLR).
  Arms: Control Group

SUMMARY:
Lumbosacral radiculopathy (LR) is among most common disorder caused due to irritation or compression of nerve pathway leading to symptoms of pain, numbness and tingling sensations along the nerve root. Lumbosacral radiculopathy consists at any lumbar region including L1-S1. Occurrence rate of Lumbosacral radiculopathy is 3-5% distributed equally in men and women affecting more men than women. It commonly occurs in late 40s in men and late 50s-60s in females. Men are more prone to develop lumbosacral radiculopathy due to mechanical disturbance during routine work.

DETAILED DESCRIPTION:
* William flexion exercises: Exercises for strengthening of gluteal and abdominal muscles which help to reduce pressure on the nerve root by promoting flexion at lumber spine such as knee to chest, double knee to chest, bridging(Gluets bridge), and straight leg raise (SLR).
* Mckenzie extension exercises: The exercises used to create space between under lying structures of lumber spine which help centralization of pain and can be performed in prone lying such as prone press ups, prone on elbow, and head lift in prone

A randomized controlled trial.

Group 1 Group 2 55 patients 55 patients

Standard treatment:

TENS (4-pole) + Hot pack for 15 minutes Standard treatment:

TENS (4-pole) + Hot pack for 15 minutes

New Intervention:

Mckenzie Extension

* Prone press-ups
* Head life in prone
* Prone on elbow
* Prone on hands
* Prone on pillow New Intervention:

William Flexion

* Single knee to chest
* Double knee to chest
* Straight Leg Raise
* Bridging
* Pelvic tilt

Each exercise will be repeated 5 minutes with 10 seconds hold and 5 sec rest. The duration of intervention will be four weeks, 3 sessions a week on alternate days and total of 12 sessions will be given. Data will be collected in three phases Pre-Treatment at end of second week and at the completion of treatment time i.e end of 4th week.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females with age between 40-60 years

  * Patients referred from neuro and orthopedic departments with diagnosed lumbosacral radiculopathy.
  * Complaint of low back pain on walk, bending and after long sitting with positive slump test.
  * Complaint of low back pain, and numbness and tingling in leg with positive SLR test

Exclusion Criteria:

* • Lumbar Trauma

  * Any other orthopedic and neurological conditions of hip and lumbosacral spine.
  * Hip Fracture
  * Malignancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-01-21 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  0 means no pain and 10 means worst pain ever felt
Flexi curve ruler | 4 weeks
  to measure the lumber cure
Bubble inclinometer | 4 weeks
  Measure the cure
King Health Questionnaire quality of life | 4 weeks
  lesser score means low quality of life and higher score means better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Isra niversity, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No